CLINICAL TRIAL: NCT00495391
Title: Phase II, Randomized, Double-blind, Placebo-controlled Study of Nitazoxanide in Combination With Peginterferon Alfa-2a and Ribavirin in Patients With Hepatitis C Who Have Failed to Respond to a Prior Course of Peginterferon and Ribavirin
Brief Title: Study of Nitazoxanide, Peginterferon Alfa-2a and Ribavirin for the Treatment of Hepatitis C
Acronym: STEALTHC-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM01-2025
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — nitazoxanide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral 500 mg nitazoxanide twice daily for 4 weeks followed by oral 500 mg nitazoxanide twice daily plus weekly injections of peginterferon alfa-2a plus oral ribavirin (1000 mg if <75 kg body weight or 1200 mg if ≥75 kg body weight) in daily divided doses for 48 weeks.
  Interventions: Drug: Nitazoxanide; Biological: Peginterferon alfa-2a; Drug: Ribavirin
- 2 (Placebo Comparator): Oral placebo twice daily for 4 weeks followed by oral placebo twice daily plus weekly injections of peginterferon alfa-2a plus oral ribavirin (1000 mg if <75 kg body weight or 1200 mg if ≥75 kg body weight) in daily divided doses for 48 weeks.
  Interventions: Drug: Placebo; Biological: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Nitazoxanide — One oral 500 mg nitazoxanide tablet twice daily for 52 weeks.
  Other Names: Alinia
  Arms: 1
Drug: Placebo — One oral placebo tablet twice daily for 52 weeks.
  Arms: 2
Biological: Peginterferon alfa-2a — Weekly injections of 180µg peginterferon alfa-2a for 48 weeks.
  Other Names: PEGASYS
Drug: Ribavirin — 1000 mg (if <75 kg body weight) or 1200 mg (if ≥75 kg body weight) ribavirin in divided daily doses for 48 weeks.
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to determine if nitazoxanide in combination with peginterferon alfa-2a and ribavirin is safe and effective in treating chronic hepatitis C in patients that have previously failed to respond to treatment with peginterferon and ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C genotype 1.
* Failed to respond to ≥12 weeks of peginterferon and ribavirin (<2 log10 drop in Hepatitis C Virus Ribonucleic Acid (HCV RNA) at week 12 or detectable Hepatitis C Virus Ribonucleic Acid (HCV RNA) at week 24).

Exclusion Criteria:

* Females of child-bearing age who are either pregnant, breast-feeding or not using birth control and are sexually active.
* Males whose female partners are either pregnant or of child-bearing potential or not using birth control and are sexually active.
* Other causes of liver disease including autoimmune hepatitis.
* Transplant recipients receiving immune suppression therapy.
* Screening tests positive for Anti-Hepatitis A Virus Immunoglobulin M Antibody (anti-HAV IgM Ab), Hepatitis B's antigen (HBsAg), Anti-Hepatitis B core antigen Immunoglobulin M Antibody (anti-HBc IgM Ab) or Anti-Human Immunodeficiency Virus Antibody (anti-HIV Ab).
* Decompensated cirrhosis, history of variceal bleeding, ascites, hepatic encephalopathy, Child-Turcotte-Pugh (CTP) score >6 or Model for End-stage Liver Disease (MELD) score >8.
* Alcohol consumption of >40 grams per day or an alcohol use pattern that will interfere with the study.
* Absolute neutrophil count <1500 cells/mm3; platelet count <135,000 cells/mm3; hemoglobin <12 g/dL for women and <13 g/dL for men; or serum creatinine concentration ≥1.5 times Upper Limit of Normal (ULN).
* Hypothyroidism or hyperthyroidism not effectively treated with medication.
* Hemoglobin A1C (HgbA1c) >7.5 or history of diabetes mellitus.
* Body Mass Index (BMI) >28.
* History or other clinical evidence of significant or unstable cardiac disease.
* History or other clinical evidence of chronic pulmonary disease associated with functional impairment.
* Serious or severe bacterial infection(s).
* Ulcerative or hemorrhagic/ischemic colitis.
* Pancreatitis.
* History of severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization.
* History of uncontrolled severe seizure disorder.
* Requires concomitant theophylline or methadone.
* History of immunologically mediated disease requiring more than intermittent anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids.
* History or other evidence of severe retinopathy or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension.
* Hemoglobinopathies.
* History of hypersensitivity or intolerance to nitazoxanide or any of the excipients comprising the nitazoxanide tablets, peginterferon alfa-2a injectable solution or ribavirin tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Nelson, MD, Principal Investigator — University of Florida Hepatology; Stephen Harrison, MD, Principal Investigator — Brooke Army Medical Center; Arthur Berman, DO, Principal Investigator — Florida Center for Gastroenterology; Ronald Pruitt, MD, Principal Investigator — Nashville Medical Research Institute; Ahmed Aijaz, MD, Principal Investigator — Stanford University; Ramsey Cheung, MD, Principal Investigator — VA Palo Alto Health Care System; Ira Jacobson, MD, Principal Investigator — Weill Medical College of Cornell University; Mitchell Shiffman, MD, Principal Investigator — McGuire VA Medical Center; Joseph Lim, MD, Principal Investigator — Yale University Digestive Diseases; Norman Gitlin, MD, Principal Investigator — Atlanta Gastroenterology Associates
Locations (10):
- United States (10):
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Stanford University School of Medicine, Stanford, California
  - Yale University Digestive Diseases, New Haven, Connecticut
  - University of Florida Hepatology, Gainesville, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Weill Cornell Medical College, New York, New York
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - McGuire VA Medical Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients from 10 study sites in the United States, including a Veterans Administrations hospital.
Groups:
- NTZ+PR: Oral 500 mg nitazoxanide twice daily for 4 weeks followed by oral 500 mg nitazoxanide twice daily plus weekly injections of peginterferon alfa-2a plus oral ribavirin (1000 mg if <75 kg body weight or 1200 mg if ≥75 kg body weight) in daily divided doses for 48 weeks.
  Ribavirin : 1000 mg (if <75 kg body weight) or 1200 mg (if ≥75 kg body weight) ribavirin in divided daily doses for 48 weeks.
  Nitazoxanide : One oral 500 mg nitazoxanide tablet twice daily for 52 weeks.
  Peginterferon alfa-2a : Weekly injections of 180µg peginterferon alfa-2a for 48 weeks.
- Placebo+PR: Oral placebo twice daily for 4 weeks followed by oral placebo twice daily plus weekly injections of peginterferon alfa-2a plus oral ribavirin (1000 mg if <75 kg body weight or 1200 mg if ≥75 kg body weight) in daily divided doses for 48 weeks.
  Ribavirin : 1000 mg (if <75 kg body weight) or 1200 mg (if ≥75 kg body weight) ribavirin in divided daily doses for 48 weeks.
  Peginterferon alfa-2a : Weekly injections of 180µg peginterferon alfa-2a for 48 weeks.
  Placebo : One oral placebo tablet twice daily for 52 weeks.
Period: Overall Study
Arm/Group | NTZ+PR | Placebo+PR
Started | 42 | 22
From Baseline to Week 8 | 31 | 20
From Baseline to Week 16 | 24 | 11
From Baseline to End of Treatment | 6 | 1
From Baseline to End of Follow up | 6 | 1
Completed | 6 | 1
Not Completed | 36 | 21
Not completed — Lack of Efficacy | 34 | 18
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NTZ+PR | Placebo+PR | Total
Number analyzed (Participants) | 42 | 22 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 21 | 60
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8) | 53 (6) | 53.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 29 | 14 | 43
Region of Enrollment [Number; unit: participants]
  United States | 42 | 22 | 64

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection 24 weeks after the end of treatment. All others were considered non-responders.
Time Frame: 24 weeks after end of treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 42 | 22
participants
  Responders | 3 | 0
  Non-responders | 39 | 22

2. Secondary Outcome: End of Treatment Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection at the end of treatment. All others were considered non-responders.
Time Frame: At end of treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 42 | 22
participants
  Responders | 6 | 1
  Non-responders | 36 | 21

3. Secondary Outcome: Early Virologic Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection after 12 weeks of combination therapy.
Time Frame: After 12 weeks combination treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 42 | 22
participants
  Responders | 3 | 0
  Non-responders | 39 | 22

4. Secondary Outcome: Rapid Virologic Response (HCV RNA Below Lower Limit of Detection)
Description: Hepatitis C Virus Ribonucleic Acid (HCV RNA) below lower limit of detection after 4 weeks of combination therapy.
Time Frame: After 4 weeks combination treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 42 | 22
participants
  Responders | 2 | 0
  Non-responders | 40 | 22

5. Secondary Outcome: Changes in ALT
Description: This analysis was conducted using a comparison of changes in Alanine aminotransferase (ALT) from baseline through week 8, week 16, end of treatment and end of follow up.
Time Frame: From baseline to week 8
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 31 | 20
participants
  Remains Elevated | 14 | 8
  Elevated to Normal | 7 | 2
  Remains Normal | 9 | 9
  Normal to Elevated | 1 | 1

6. Secondary Outcome: Changes in ALT
Description: as for outcome 5
Time Frame: From baseline to week 16
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 24 | 11
participants
  Remains Elevated | 6 | 2
  Elevated to Normal | 6 | 2
  Remains Normal | 12 | 6
  Normal to Elevated | 0 | 1

7. Secondary Outcome: Changes in ALT
Description: as for outcome 5
Time Frame: From baseline to end of treatment
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 6 | 1
participants
  Remains Elevated | 0 | 0
  Elevated to Normal | 1 | 0
  Remains Normal | 5 | 1
  Normal to Elevated | 0 | 0

8. Secondary Outcome: Changes in ALT
Description: as for outcome 5
Time Frame: From baseline to end of follow up
Measure: Number; unit: participants
Arm/Group | NTZ+PR | Placebo+PR
Number analyzed (Participants) | 6 | 1
participants
  Remains Elevated | 0 | 0
  Elevated to Normal | 1 | 0
  Remains Normal | 4 | 1
  Normal to Elevated | 1 | 0

ADVERSE EVENTS:
Time Frame: 2 years, 1 month
Arm/Group | NTZ+PR | Placebo+PR
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/22
Other Adverse Events (participants affected / at risk) | 42/42 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTZ+PR (N=42) | Placebo+PR (N=22)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney Calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Edema Larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTZ+PR (N=42) | Placebo+PR (N=22)
Asthenia (General disorders) | 23 (23) | 10 (10)
Pain Abdo (Gastrointestinal disorders) | 9 (9) | 2 (2)
Headache (General disorders) | 9 (9) | 6 (6)
Pain Back (General disorders) | 6 (6) | 0 (0)
Flu Synd (General disorders) | 5 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 17 (17) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (10) | 4 (4)
Anorexia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Constip (Gastrointestinal disorders) | 5 (5) | 2 (2)
Liver Func Abnorm (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 20 (20) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (12) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 11 (11) | 5 (5)
Agitation (Nervous system disorders) | 12 (12) | 6 (6)
Depression (Nervous system disorders) | 8 (8) | 5 (5)
Insomnia (Nervous system disorders) | 8 (8) | 4 (4)
Anxiety (Nervous system disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (5)
Skin Dry (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Cough Inc (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Albuminuria (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Cramps Leg (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Polyuria (Renal and urinary disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Presentation and/or publication is encouraged provided the Sponsor is notified in advance and given the opportunity to review the manuscript or abstract 30 days prior to its submission for presentation at a scientific meeting or for publication in a scientific journal. The investigators will have complete autonomy regarding the content and wording including the decision of whether or not to publish.